CLINICAL TRIAL: NCT06245759
Title: Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, China
Brief Title: The Prognostic Impact of Tumor Location in Non-Muscle-Invasive Bladder Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Lilong Liu, Director, Huazhong University of Science and Technology
Other Study IDs: TJIRB20230888
Record Dates: First submitted 2024-01-23; First posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-01

CONDITIONS: Non-Muscle-Invasive Bladder Cancer; Bladder Cancer
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- the U.S. National Cancer Center SEER database: The Chinese NMIBC cohort includes patients from January 1996 to December 2019 at 15 institutions.
  Interventions: Other: This was a retrospective study and no patient intervention was performed
- the Chinese Bladder Cancer Alliance CBCC database: SEER*Stat software (version 8.4.1.1) collected 17 registries cohort data on NMIBC patients diagnosed between 2000 and 2020.
  Interventions: Other: This was a retrospective study and no patient intervention was performed

INTERVENTIONS:
Other: This was a retrospective study and no patient intervention was performed — This was a retrospective study and no patient intervention was performed

SUMMARY:
Based on large sample size studies at home and abroad, the prognosis of patients with non-muscular invasive bladder cancer in different sites undergoing transurethral bladder tumor resection was determined, providing important guidance for subsequent clinical treatment and surgical instrument development.

DETAILED DESCRIPTION:
Background Most bladder cancers are non-muscle invasive bladder cancer (NMIBC), and transurethral resection of bladder tumors (TURBT) is the standard treatment. However, postoperative recurrence poses a challenge, and the influence of bladder tumor location on prognosis is unclear. This study aims to investigate how tumor location affects NMIBC patients' prognosis undergoing TURBT, and seeks optimal surgical approaches.

Methods Conducted a multicenter study, including Chinese NMIBC data from 15 hospitals (1996-2019) and SEER 17 registries (2000-2020). Analyzed patients initially diagnosed with NMIBC undergoing TURBT or partial cystectomy, excluding cases with lost follow-up or missing data. Studied overall survival (OS), disease-specific survival (DSS), and recurrence-free survival (RFS). Employed Kaplan-Meier, Cox regression, and propensity score matching to explore the association between tumor location and prognosis. Stratified populations were analyzed to minimize bias.

Findings This study, involving 118,477 NMIBC patients, highlighted tumor location as a crucial factor impacting post-TURBT prognosis. Anterior wall and dome tumors independently predicted adverse outcomes in both cohorts. For anterior wall tumors, Chinese cohort showed OS HR 4.35, p < 0.0001; RFS HR 2.21, p < 0.0001; SEER OS HR 1.10, p = 0.0001; DSS HR 1.13, p = 0.0183. Dome tumors displayed similar trends (Chinese NMIBC cohort OS HR 7.91, p < 0.0001; RFS HR 2.12, p < 0.0001; SEER OS HR 1.05, p = 0.0087; DSS HR 1.14, p = 0.0006). Partial cystectomy significantly improved dome tumor survival compared to standard TURBT (p < 0.01).

Interpretation This study reveal that NMIBC tumor location significantly influences TURBT treatment outcomes. Specifically, tumors in the anterior wall and bladder dome have worse post-TURBT prognosis. Compared to TURBT, partial cystectomy improves prognosis for bladder dome tumors. This study guides personalized treatment and prognosis management for NMIBC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Initially diagnosed with non-muscular invasive bladder cancer (NMIBC) who underwent TURBT or partial cystectomy.
2. The follow-up data of the patients were complete.
3. The tumor location information were complete.

Exclusion Criteria:

1. Patients with unknown survival time or missing tumor location information were excluded.
2. Exclude patients with missing pathological results.
3. Exclude patients who have had TURBT before.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study utilized the Chinese NMIBC cohort as well as the SEER 17 registries cohort for its investigation. The Chinese NMIBC cohort contains data of patients between January 1996 and December 2019, at 14 institutions. SEER*Stat software (version 8.4.1.1) was used for collecting 17 registries cohort data on patients diagnosed with NMIBC between 2000 and 2020.
Sampling Method: Non-Probability Sample
Enrollment: 120000 (Estimated)
Dates: Start 2023-08-31 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival time | up to 20 years
  OS, defined as the time from the first diagnosis to death from any cause or the last follow-up for surviving patients
Recurrence free survival time | up to 16 years
  Recurrence-free survival (RFS) is the time from the time a patient achieved complete response after antineoplastic therapy to the time of recurrence or the end of follow-up. The longer the relapse-free survival time, the better the efficacy of anti-tumor therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Ke Chen, MD/PhD, Study Chair — Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, China
Locations (1):
- Ke Chen, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu L, Li K, Wang SG, Wang J, Yao Z, Xie Y, Ji Z, Chen Z, Hu H, Chen H, Hu J, Hou Y, Liu Z, Li Y, Ding Y, Kuang Y, Xun Y, Hu J, Zhang J, Li H, Chong T, Bi J, Wang Z, Wang Y, Zhang P, Wei Q, Chen Z, Li L, Huang J, Liu Z, Chen K; Chinese Bladder Cancer Consortium. The prognostic impact of tumor location in nonmuscle-invasive bladder cancer patients undergoing transurethral resection: insights from a cohort study utilizing Chinese multicenter and SEER registries. Int J Surg. 2024 Sep 1;110(9):5641-5651. doi: 10.1097/JS9.0000000000001675. PMID 38788195